CLINICAL TRIAL: NCT06896292
Title: Efficacy, Feasibility, and Acceptability of a Hybrid Patient Care Model in Improving Access to Guideline Recommended Antenatal Preventive Care
Brief Title: Testing a Digital Tool to Support Healthy Pregnancies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter and New England Health (Other)
Responsible Party: Principal Investigator, Dr Melanie Kingsland, Program Manager, Hunter and New England Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025/ETH00079
Record Dates: First submitted 2025-03-13; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Preventive Behaviors; Antenatal Care and Delivery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data collection staff that are involved in undertaking telephone interviews with control and intervention group participants will not be aware of their group allocation when collecting data for primary outcome measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hybrid care model (Experimental): The Hybrid care model will involve guideline-recommended preventive care (AAH) for smoking, nutrition, alcohol, physical activity and gestational weight gain- standard care as it is currently delivered within antenatal appointments conducted by maternity services + use of a digital support tool. The digital tool will allow patients to undertake self-assessment of smoking, nutrition, alcohol, physical activity and gestational weight gain risks, receive information and make self-referrals to support services at a time and in a way that suits them. Self-assessment results and information on self-referrals will be provided to antenatal clinicians prior to appointments to support clinician follow-up. The provision of preventive care via the digital support tool will facilitate more streamlined appointments by addressing priority issues and freeing up appointment time to address issues most relevant to the participant.
  Interventions: Behavioral: Hybrid care model
- Usual care model (Active Comparator): Usual guideline-recommended preventive care (AAH) for smoking, nutrition, alcohol, physical activity and gestational weight gain- standard care as it is currently delivered within antenatal appointments conducted by maternity services
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Hybrid care model — Participants will receive usual antenatal care (in-person), plus the digital support tool. A co-design process was used to develop the tool based on consumer feedback.
  The tool is based on the recommended Assess/ask, Advise, Help approach to preventive care for smoking, nutrition, alcohol, physical activity and gestational weight gain.
  Participants will be prompted (via SMS) to use the digital support tool at regular intervals throughout their pregnancy to self-assess health risks and be reminded of recommendations and available coaching services.
  Arms: Hybrid care model
Other: Usual Care — Participants will receive usual antenatal care (in-person), which is recommended to include the delivery of preventive care using the AAH model for smoking, nutrition, alcohol, physical activity and gestational weight gain.
  Arms: Usual care model

SUMMARY:
The delivery of preventive care for modifiable health risks (smoking, nutrition, alcohol, physical activity and gestational weight gain) is a critical part of antenatal care. Clinical guidelines recommend that preventive care is delivered using three elements: Ask, Advise, and Help (AAH). Unfortunately, the AAH model for modifiable risk factors is not routinely delivered to all pregnant people in face-to-face antenatal visits. We will test if adding a digital support tool to usual antenatal care increases the provision of guideline-recommended preventive care for smoking, nutrition, alcohol, physical activity and gestational weight gain, compared to usual antenatal care at two maternity services based at Maitland Hospital and Manning Base Hospital in New South Wales, Australia. The digital support tool will provide the opportunity for pregnant people to self-assess smoking, nutrition, alcohol, physical activity and gestational weight gain risk prior to their antenatal visits, while also being provided with tailored guideline-based information and the opportunity to self-refer to support services. Use of the digital support tool may also prompt pregnant people and/or their antenatal clinicians to have discussions around smoking, nutrition, alcohol, physical activity and gestational weight gain risks at antenatal appointments. As well as assessing impact on receipt of care for smoking, nutrition, alcohol, physical activity and gestational weight gain, we will also explore the feasibility, acceptability, barriers/enablers to use and content and functional preferences of the digital support tool for pregnant people.

ELIGIBILITY:
Inclusion Criteria:

* Any pregnant person (aged 18 years and over) with a scheduled first antenatal appointment at one of the two participating maternity services
* Sufficient level of English language proficiency to access and use the digital support tool and complete follow-up surveys.

Exclusion Criteria:

* Any pregnant person who has had an adverse pregnancy outcome. As per previous studies undertaken by the research team, this criterion will be assessed by review of relevant medical record fields and anyone who meets this criterion will be flagged to exclude from invitation to the study or from being included in any trial related data collection or contacts.
* No registered mobile phone number

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Receipt of preventive care (Assessment of health risks) | Throughout study via digital tool analytics and during interviews conducted approximately 1-3 weeks following three antenatal appointments, that is, the first appointment (14-20 weeks), 28-week and 36-week gestation appointment.
  The percentage of pregnant people (N=840) receiving assessment of all health risks (smoking, nutrition, alcohol, physical activity and gestational weight gain) via the digital support tool or their antenatal provider.
Receipt of preventive care (Advice about health risks) | Throughout study via digital tool analytics and during interviews conducted approximately 1-3 weeks following three antenatal appointments, that is, the first appointment (14-20 weeks), 28-week and 36-week gestation appointment.
  The percentage of pregnant people (N=840) receiving advice on all relevant health risks (smoking, nutrition, alcohol, physical activity and gestational weight gain) via the digital support tool or their antenatal provider.
Receipt of preventive care (Help to address health risks) | Throughout study via digital tool analytics and during interviews conducted approximately 1-3 weeks following three antenatal appointments, that is, the first appointment (14-20 weeks), 28-week and 36-week gestation appointment.
  The percentage of pregnant people (N=840) who are referred to at least one preventive health service for an identified health risk (clinician referral or self-referral) via the digital support tool or their antenatal provider.

OTHER OUTCOMES:
Process Measures | Throughout study via digital tool analytics and during interviews conducted approximately 1-3 weeks following three antenatal appointments, that is, the first appointment (14-20 weeks), 28-week and 36-week gestation appointment.
  We will collect a range of process measures to better understand acceptability and participant preferences for the digital support tool. Process measures have been informed by the Design and Evaluation Framework for Digital Health Interventions. We will assess:
  * use/adoption
  * barriers
  * enablers
  * acceptability
  * preferences (content and function)

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Maitland Hospital Maternity Services, Maitland, New South Wales
  - Manning Hospital Maternity Services, Taree, New South Wales

IPD SHARING:
Plan to Share IPD: Yes
If data is requested by other researchers following the publication of study results, a reasonable request in writing to the Chief Investigator (Dr Kingsland) will be required. Only deidentified data will be provided. Ongoing custody of the data will remain with the Chief Investigator- Dr Kingsland.